CLINICAL TRIAL: NCT03470402
Title: Decision Support for BRCA Testing in Ethnically Diverse Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR3676
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; BRCA1 Mutation; BRCA2 Mutation; Ovarian Cancer
Keywords: Breast Cancer Prevention; Genetic Testing; Genetic Counseling; Personalized Prevention; Precision Prevention; Precision Medicine; Risk Assessment; Decision Making; Decision Aid
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: A cluster randomization in which both a provider and his/her enrolled patients will be enrolled in either the intervention or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Women who screen as eligible for BRCA genetic counseling will receive the education and decision support tool, RealRisks, along with standard educational material and a high-risk message. The high-risk status of the women will also be flagged in the online tool used by the hospital to visualize electronic health record data (iNYP).
  The enrolled health care providers of these women will be given access to BNAV, which summarizes their enrolled patients' breast cancer risk profiles and provides educational resources on genetic testing and prevention options. Before their clinical encounter with an enrolled patient, these providers will also be sent the personalized breast cancer risk summary that is created by data the patient entered into RealRisks.
  Interventions: Other: RealRisks; Other: BNAV; Other: iNYP; Other: Standard Educational Material; Other: High-Risk Message
- Control group (Active Comparator): Women who screen as eligible for BRCA genetic counseling will receive standard educational material and a high-risk message. The high-risk status of the women will also be flagged in the online tool used by the hospital to visualize electronic health record data (iNYP).
  Interventions: Other: iNYP; Other: Standard Educational Material; Other: High-Risk Message

INTERVENTIONS:
Other: RealRisks — RealRisks is a web-based patient decision aid with modules on risk assessment, family history and breast cancer, genetic testing, and prevention options. Participants enter family history data into RealRisks, and RealRisks calculates 5-year breast cancer risk, lifetime breast cancer risk, and the probability of carrying a BRCA mutation. This information is then interactively presented to the participant. RealRisks facilitates the participant in identifying their intention to undergo BRCA genetic testing and the factors that are important to the participant in making this decision. RealRisks produces a summary of all of this information that the participant can print and take with her to a health care appointment.
  Other Names: RealRisks Decision Aid
  Arms: Intervention group
Other: BNAV — BNAV is a web-based decision support tool for healthcare providers with educational modules on genetic testing, chemoprevention, patient-centered care, and screening. BNAV also provides providers with a table outlining their enrolled patients' breast cancer risk, eligibility for genetic testing, and stated preferences.
  Other Names: Breast Cancer Risk Navigation Tool; BNAV Toolbox
  Arms: Intervention group
Other: iNYP — Enrolled patients will have their eligibility for BRCA genetic testing flagged in iNYP, the hospital's portal for visualizing EHR data (standard practice).
Other: Standard Educational Material — Enrolled patient participants will be sent standard educational brochures on genes and breast cancer and the CUMC breast cancer prevention clinic
  Other Names: Standard Educational Brochures
Other: High-Risk Message — Enrolled patient participants will receive a letter that informs them that they meet eligibility criteria for BRCA genetic testing, outlines prevention options, and recommends discussing genetic counseling referral with their health care provider (standard practice).
  Other Names: High Risk Letter

SUMMARY:
The objective of this study is to expand genetic testing for hereditary breast and ovarian cancer syndrome to a broader population of high-risk women by prompting appropriate referrals from the primary care setting with the use of an electronic health record-embedded breast cancer risk navigation (BNAV) tool. To address patient-related barriers to genetic testing, the investigators developed a web-based decision aid, RealRisks, which is designed to improve genetic testing knowledge, accuracy of breast cancer risk perceptions, and self-efficacy to engage in a collaborative dialogue about genetic testing.

The study design is a randomized controlled trial of patient educational materials and provider electronic health record (EHR) notice alone (control arm) or in combination with RealRisks and BNAV (intervention arm). The investigators hypothesize that combining the patient-centered RealRisks with the provider-centered BNAV will increase appropriate uptake of genetic counseling. The investigators also hypothesize that genetic counseling decisions will be more informed, and result in less decision conflict and improved shared decision making.

DETAILED DESCRIPTION:
Hereditary breast and ovarian cancer syndrome (HBOC) is an inherited condition that is most commonly associated with mutations in the BRCA1 and BRCA2 genes. Mutation carriers have lifetime risks of breast and ovarian cancer of 60-80% and 20-40%, respectively. Risk management options include intensive breast cancer screening, risk-reducing surgeries, and chemoprevention, which have been shown to improve early detection and reduce cancer incidence and mortality. In particular, prophylactic bilateral salpingo-oophorectomy has been associated with a 60-77%reduction in all-cause mortality among BRCA mutation carriers. Based upon U.S. Preventive Services Task Force guidelines, an estimated 5%-10% of women unaffected with breast cancer are eligible for genetic testing for HBOC, but only 14% of those eligible were referred and 4% had BRCA genetic testing. Many women may be unaware of their high-risk status due to our inability to adequately screen them in the primary care setting. Other reasons for low uptake include inadequate time for counseling and insufficient knowledge about risk-reducing strategies. Women from racial/ethnic minorities are less likely to seek genetic testing for HBOC, contributing to poorer clinical outcomes in these populations compared to non-Hispanic whites. Alternatively, decreasing inappropriate genetics referrals is also important for reducing anxiety and allowing genetic services to be used more efficiently. More research is needed to develop optimal strategies for engaging high-risk women in informed decision-making about genetic testing for HBOC.

The objective of this study is to expand genetic testing for hereditary breast and ovarian cancer syndrome to a broader population of high-risk women by prompting appropriate referrals from the primary care setting with the use of an electronic health record-embedded breast cancer risk navigation (BNAV) tool. To address patient-related barriers to genetic testing, the investigators developed a web-based decision aid, RealRisks, which is designed to improve genetic testing knowledge, accuracy of breast cancer risk perceptions, and self-efficacy to engage in a collaborative dialogue about genetic testing.

The study design is a randomized controlled trial of patient educational materials and provider EHR notice alone (control arm) or in combination with RealRisks and BNAV (intervention arm). The investigators hypothesize that combining the patient-centered RealRisks with the provider-centered BNAV will increase appropriate uptake of genetic counseling. The investigators also hypothesize that genetic counseling decisions will be more informed, and result in less decision conflict and improved shared decision making.

ELIGIBILITY:
Inclusion Criteria (Patient Participants):

* Women, age 21-75 years
* Meets criteria for genetic testing based on family history
* Sees a primary care provider in the Columbia University (CUMC) /New York Presbyterian (NYP) Ambulatory Care Network
* Understands as is willing to provide informed consent in English or in Spanish

Exclusion Criteria (Patient Participants):

* Prior genetic counseling or testing for hereditary breast and ovarian cancer (HBOC)
* A personal history of breast or ovarian cancer

Inclusion Criteria (Health Care Provider Participants):

* Primary care providers, such as attending physicians, residents, nurse practitioners, physician assistants, and midwives, who see patients at CUMC/NYP Ambulatory Care Network clinics
* Able to provide informed consent

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Uptake rate of genetic counseling by 6 months | Up to 6 months
  The primary endpoint is to determine the uptake of genetic counseling for HBOC syndrome by 6 months in the intervention arm (RealRisks Decision Aid and BNAV toolbox) compared to the control arm (Standard educational materials)

SECONDARY OUTCOMES:
Change in patient decision conflict scale score | Baseline, Post Intervention/Control (1 Month), Post Clinic Encounter (Approximately 6 Weeks), 6 Months
  The decisional conflict scale (DCS) measures personal perceptions of: uncertainty in choosing options; modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and effective decision making (in full version) such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice.
  It includes 10 yes/no items (0=yes, 2=unsure, 4=no). Analysis: Item scores are summed, divided by 10, and multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict). A lower score indicates a better outcome.
Shared Decision Making (Likert Scale Score) | Post Clinic Encounter (Approximately 6 Weeks)
  The Shared Decision Making (SDM) questionnaire collects information on the process in which clinicians and patients work together to make decisions and select tests, treatments and care plans based on clinical evidence that balances risks and expected outcomes with patient preferences and values. It consists of 9 items with each item scored on a 6-point Likert scale (0=completely disagree to 5=Complete Agree) from the SDM-Q-9.
  Analysis: A raw total score between 0 and 45 calculated by summing the scores of all items. If required, imputation of up to two missing items using the mean of the items that made up the raw score. For the standardization of the raw score, a linear transformation into a scale ranging from 0 to 100 (multiplication of the raw score by 20/9), with zero indicating the lowest level of perceived SDM and 100 indicating the highest level of perceived SDM (better outcome).
Patient Informed Choice Score | 6 Months
  The degree to which a decision is based on relevant, good quality information, and reflects the decision-maker's values. To compare between the intervention and control group at 6 months. To be an informed choice, a patient needs a good knowledge score and a decision that is consistent with their attitude score. Analysis: Informed Choice= Good knowledge (score 50% and above) AND Positive Attitude (score 22 and above) AND positive decision ("I decided to get genetic testing" or "I was already tested"), OR Good knowledge AND Negative attitude (score 21 and below) AND negative decision ("I decided not to get genetic testing") Uninformed Choice: Poor knowledge, OR Good knowledge, but uptake inconsistent with attitudes Analysis: Uninformed Choice= Good knowledge (score 50% and above) AND Negative attitude AND positive decision OR Good knowledge AND Negative Attitude Score AND positive decision, OR Poor knowledge (49% and below).

OTHER OUTCOMES:
Change in Risk Perceptions (Likert Scale Score) | Baseline, Post Intervention/Control (1 Month), Post Clinic Encounter (Approximately 6 Weeks), 6 Months
  Change in the accuracy of risk perception among patient participants. Perception will be assessed by comparing a patients perceived risk with their actual risk, and to compare between intervention and control group will be assessed at baseline, after receiving intervention or control materials, after the clinic encounter, and at 6 months. Perceived risk will be measured by Likert and numerical scales and actual risk will be determined by a model.
  Likert Scale: Eight 6-point items measuring perceived ability to perform mathematical tasks and preferences for receiving word-based or number-based information.
  Analysis: Question 7 reverse coded, then find mean of all 8 item scores. Score 1 = least accurate risk perception, Score 6= most accurate risk perception. A higher score indicates a better outcome.
Change in Breast Cancer Worry (Likert Scale Score) | Baseline, Post Intervention/Control (1 Month), Post Clinic Encounter (Approximately 6 Weeks), 6 Months
  Likert Scale measuring breast cancer worry among patient participants. To compare between intervention and control group at baseline, after receiving intervention or control materials, after the clinic encounter, and at 6 months Two 7-point items measuring how often patient worries about developing cancer and how much this worry interferes with everyday life. 1="none of the time"; 4="Some of the time"; 7="All of the time". Scores summed.Higher score indicates more worry and more interference with everyday life. Lower score indicates a better outcome.
Change in Breast Cancer Knowledge scale score | Baseline, Post Intervention/Control (1 Month), Post Clinic Encounter (Approximately 6 Weeks), 6 Months
  True false scale measuring knowledge of breast cancer and HBOC among patient participants. To compare between intervention and control group at baseline, after receiving intervention or control materials, after the clinic encounter, and at 6 months 11 true/false items Analysis: Sum # correct; 50%-100% correct is considered good knowledge and indicates better outcome, 0-49% correct is considered poor knowledge.
Change in Attitudes (Likert Scale Score) | Baseline, Post Intervention/Control (1 Month), Post Clinic Encounter (Approximately 6 Weeks), 6 Months
  Likert scale measuring patient attitudes towards BRCA genetic testing. To compare between intervention and control group at baseline, after receiving intervention or control materials, after the clinic encounter, and at 6 months Four 7-point Likert scale items, which are summed; 22 as cut-point for positive/negative items. 22 and above considered positive attitudes. A positive attitude is indicative of a better outcome. 21 and below considered negative attitudes. Up to one missing item will be imputed using the average of the remaining three item scores.
Change in Decision Self Efficacy (Likert Scale Score) | Baseline, Post Intervention/Control (1 Month), 6 Months
  Likert scale measuring degree of self efficacy in making a genetic testing decision among patient participants. To compare between intervention and control group at baseline, after receiving intervention or control materials, after the clinic encounter, and at 6 months 11 5-point Likert scale items (0=not at all confident - 4=very confident) Analysis: items are summed, divided by 11, and multiplied by 25. Scores range from 0 (extremely low efficacy) to 100 (extremely high efficacy). A higher score indicates a better outcome.
Change in Decision Regret (Likert Scale Score) | Post Clinic Encounter (Approximately 6 Weeks), 6 months
  Likert scale measuring measuring the extent to which a patient regrets the decision to undergo or not undergo genetic counseling. To compare between intervention and control groups after the clinic encounter and at 6 months Low-literacy option: five 5-point Likert scale items (1=Strongly Agree - 5=Strongly Disagree) measuring whether regret was felt to be present, whether the decision was the right one, whether the patient would make the same decision again, whether the decision was a wise one, and whether the decision had resulted in harm.
  Analysis: Reverse code Regret_2 and Regret_4. Subtract 1 from each item score and multiply by 25. Mean scores of items Regret_1-Regret_5; A score of 0 means no regret, while a score of 100 means high regret. A lower score indicates a better outcome.
Change in Confidence in Managing Patients with a Family History of Breast/Ovarian Cancer (Likert Scale Score) | Baseline, 6 Months
  Likert scale measuring confidence in managing patients with a family history of breast/ovarian cancer among health care provider participants. To compare between intervention and control group at baseline and six months Three questions ascertaining respondents' perceived level of confidence in their knowledge of medical statistics, ability to effectively communicate medical statistics to patients and/or families, and ability to help patients and/or families understand information about probabilities or risks.
  6-point Likert scale: "Not at all" to "Extremely" confident. Analysis: mean scores, 0= "Not at all" confident - 5= "Extremely" Confident. A higher score indicates a better outcome.
Change in Provider Knowledge questionnaire score | Baseline, 6 Months
  Three "Agree/Disagree" statement and two multiple choice questions measuring BRCA genetic testing knowledge among health care provider participants. To compare between intervention and control group at baseline and 6 months.
  Analysis: Number of multiple choice items answered correctly ( 0, 1, or 2 items answered correctly). Score range from 0-2. The higher the score, the greater the provider knowledge. A higher score indicates a better outcome.
Change in Provider Attitudes | Baseline, 6 Months
  Likert scale measuring attitudes held by health care provider participants regarding BRCA genetic testing. To compare between intervention and control group at baseline and 6 months.
  One statement, 7 point Likert scale: 0="strongly disagree" - 6= "strongly agree" Analysis: High scores indicate stronger intention, perception of stronger social pressure, and perception of greater control. A higher score indicates a better outcome.
Change in Orientation Towards Shared Decision Making (Likert Scale Score) | Baseline, 6 Months
  Likert scale measuring the extent to which a respondent believes that patients desire information and should be part of decision making process. Among health care provider participants. To compare between intervention and control group at baseline and 6 months.
  9-item scale measuring the extent to which a respondent believes that patients desire information and should be part of the decision making process.
  6-point Likert Scale: 0= "Strongly Disagree" - 5= "Strongly Agree" Analysis: Total score, score ranging from 0-45, lower score= patient centered, higher score= doctor-centered. The greater the change in orientation towards shared decision making, the better the outcome.
Change in Subjective Norms | Baseline, 6 Months
  Likert scale measuring extent to which providers believe others would expect them to refer patients to BRCA genetic testing. For health care provider participants. To compare between intervention and control group at baseline and 6 months.
  7 point item: 0= "Strongly disagree" - 6= "Strongly agree" Analysis: High scores indicate perception of stronger social pressure and indicates a better outcome.
Change in Perceived behavioral control | Baseline, 6 Months
  Likert scale measuring extent to which providers believe they are able to refer patients to BRCA genetic testing. For provider participants. To compare between intervention and control group at baseline and 6 months.
  7 point item: 0= "very difficult" - 6 = "very easy" Analysis: High scores indicate perception of greater control. A higher score indicates a better outcome.
Change in behavior Intention test score | Baseline, 6 Months
  Multiple choice measuring a providers intention to refer a patient to BRCA genetic testing. For health care provider participants. To compare between intervention and control group at baseline and 6 months.
  7 point item: e.g. 0= very difficult - 6= very easy Analysis: High scores indicate stronger intention and better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Kukafka, DrPH, MA, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kukafka R, Pan S, Silverman T, Zhang T, Chung WK, Terry MB, Fleck E, Younge RG, Trivedi MS, McGuinness JE, He T, Dimond J, Crew KD. Patient and Clinician Decision Support to Increase Genetic Counseling for Hereditary Breast and Ovarian Cancer Syndrome in Primary Care: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2222092. doi: 10.1001/jamanetworkopen.2022.22092. PMID 35849397
- [Derived] Silverman TB, Vanegas A, Marte A, Mata J, Sin M, Ramirez JCR, Tsai WY, Crew KD, Kukafka R. Study protocol: a cluster randomized controlled trial of web-based decision support tools for increasing BRCA1/2 genetic counseling referral in primary care. BMC Health Serv Res. 2018 Aug 13;18(1):633. doi: 10.1186/s12913-018-3442-x. PMID 30103738